CLINICAL TRIAL: NCT02904512
Title: Inpatient Diabetes Mellitus (DM) Management With Continuous Glucose Monitoring Devices, a Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Ilias Spanakis, MD, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00070039
Record Dates: First submitted 2016-08-30; First posted 2016-09-19 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring; Surgical Instruments; Point-of-Care Systems; Blood Glucose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Continuous glucose Monitoring and Point of Care blood glucose (Active Comparator): Hospitalized patients with Diabetes Mellitus type 2 (DM2) managed with Continuous glucose monitoring (CGM) and Point of Care (POC) Finger sticks blood glucose
  Interventions: Device: Continuous glucose Monitoring (CGM) device and Point of Care (POC) blood glucose
- Point of Care (POC) blood glucose (Placebo Comparator): Hospitalized Diabetes Mellitus type 2 (DM2) patients managed with Point of Care (POC) blood glucose only
  Interventions: Other: Point of Care (POC) blood glucose

INTERVENTIONS:
Device: Continuous glucose Monitoring (CGM) device and Point of Care (POC) blood glucose — Testing Blood Glucose levels with Continuous glucose Monitoring (CGM) device and Point of Care (POC) blood glucose
  Arms: Continuous glucose Monitoring and Point of Care blood glucose
Other: Point of Care (POC) blood glucose — Testing Blood Glucose levels with Point of Care (POC) blood glucose
  Arms: Point of Care (POC) blood glucose

SUMMARY:
Several observational studies have shown that uncontrolled hyperglycemia in hospitalized patients in the non-critical care, non-Intensive Care Unit (non-ICU) setting is associated with prolonged length of stay, increased mortality and an increased incidence of infections. Randomized clinical trials in both the critical and the non-ICU settings have shown that by improving glucose control there is a decrease in the incidence of infections, length of stay and inpatient health care costs.

Continuous glucose monitoring (CGM) systems have evolved as useful devices providing excellent clinical care in patients with Diabetes Mellitus (DM). These systems detect glucose in subcutaneous interstitial fluid using a glucose sensor that transmits glucose measurements to a receiving device that reads out average glucose levels every couple of minutes.

In this clinical trial the investigators propose to examine the clinical use of CGM in hospitalized patients with Diabetes Mellitus type 2 (DM2). CGM use may improve glucometric values and clinical outcomes in hospitalized individuals with Diabetes Mellitus type 2 (DM2).

We use CGM devices to monitor but also to transmit glucose values wirelessly to monitoring devices that are in the nursing station. Half of the participants are placed on Real Time CGM (alarms turned on) and half of them are placed on blinded CGM values (alarms turned off). Nursing staff will be notified when glucose is <85 mg/dl , in order to treat and potentially prevent a potential hypoglycemic episode.

ELIGIBILITY:
Inclusion Criteria:

* History of Diabetes Mellitus type 2 (DM2) on insulin

Exclusion Criteria

* Patients that are expected to require a hospital stay ≤3 days
* Pregnant patients
* Subjects that have significant hyperglycemia or Diabetic Ketoacidosis (DKA) that requires treatment with intravenous insulin infusion
* Patients receiving glucocorticosteroids in doses (equivalent) to ≥ 20 mg of hydrocortisone/day
* Any mental condition rendering the subject incapable of understanding the objectives and potential consequences of the study
* Patients that need hospitalization in the critical care (ICU) setting.
* History of Diabetes Mellitus type 1 (DM1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified data are going to be shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous Glucose Monitoring and Point of Care Blood Glucose | Point of Care (POC) Blood Glucose
Started | 9 | 7
Completed | 6 | 7
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Transferred to ICU | 1 | 0
Not completed — Minor Bleeding at site of device insertion | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Glucose Monitoring and Point of Care Blood Glucose | Point of Care (POC) Blood Glucose | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (6.4) | 67.9 (9.6) | 69.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.1 (9.3) | 30.9 (4.9) | 32.0 (7.1)
A1c, % [Mean (Standard Deviation); unit: % of glycated hemoglobin] | 7.6 (1.3) | 8.4 (2.4) | 8.0 (1.8)
DM duration [Mean (Standard Deviation); unit: years] | 22 (12.9) | 18.4 (6.4) | 20.2 (9.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Spent in Hyperglycemia > 180 mg/dL
Time Frame: Through study completion, during hospital stay, an average of 1 week
Measure: Mean (Standard Deviation); unit: percentage of time spent > 180mg/dL
Arm/Group | Continuous Glucose Monitoring and Point of Care Blood Glucose | Point of Care (POC) Blood Glucose
Number analyzed (Participants) | 6 | 7
percentage of time spent > 180mg/dL | 35.47 (14.71) | 35.25 (29.38)

2. Primary Outcome: Percentage of Time Spent in Significant Hyperglycemia (>300 mg/dL)
Time Frame: Through study completion, during hospital stay, an average of 1 week
Measure: Mean (Standard Deviation); unit: percent of time spent > 300mg/dL
Arm/Group | Continuous Glucose Monitoring and Point of Care Blood Glucose | Point of Care (POC) Blood Glucose
Number analyzed (Participants) | 6 | 7
percent of time spent > 300mg/dL | 3.28 (5.65) | 5.52 (12.64)

3. Primary Outcome: Number of Participants With Hypoglycemic Events (< 70mg/dL)
Time Frame: Through study completion, during hospital stay, an average of 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Glucose Monitoring and Point of Care Blood Glucose | Point of Care (POC) Blood Glucose
Number analyzed (Participants) | 6 | 7
Participants | 2 | 6

ADVERSE EVENTS:
Time Frame: Adverse events collected from the patient enrollment to the end of patient hospitalization, an average of 5 days.
Arm/Group | Continuous Glucose Monitoring and Point of Care Blood Glucose | Point of Care (POC) Blood Glucose
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 2/6 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Glucose Monitoring and Point of Care Blood Glucose (N=6) | Point of Care (POC) Blood Glucose (N=7)
Transferred to ICU (for non study-related reasons) (Infections and infestations) | 1 (1) | 0 (0) — Patient developed dry gangrene and was transferred to ICU related to osteomyelitis, not the CGM in our study.
Bleeding at site of the CGM insertion (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Minor bleeding at the site of CGM insertion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT02904512/Prot_SAP_000.pdf